CLINICAL TRIAL: NCT06913257
Title: Cost-Effectiveness Analysis of Extracorporeal Shock Wave Therapy (ESWT) Combined With Standard Rehabilitation Versus Standard Rehabilitation Alone in Managing Post-Burn Scars: A Randomized Controlled Trial With Integrated Economic Evaluation
Brief Title: Cost-Effectiveness of ESWT Plus Rehabilitation vs Rehabilitation Alone in Post-Burn Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESWT-BurnCE2025
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Participants with post-burn hypertrophic scars will be randomized into two parallel arms. Stratified randomization based on scar severity ensures balanced allocation across groups. Each participant will receive a predetermined intervention and be followed for 6 months to assess changes in both clinical parameters and economic outcomes.
Who Masked: Outcomes Assessor
Masking Description: While participants, care providers, and investigators will be aware of the intervention provided, outcome assessors and the economic evaluation team will remain blinded to group allocation to reduce bias in outcome measurement and cost data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT Plus Standard Rehabilitation (Experimental): Participants in this arm will undergo extracorporeal shock wave therapy (ESWT) in addition to receiving standard rehabilitation therapy. ESWT will be administered using a standardized protocol, with treatment sessions conducted weekly for a predetermined duration, integrated with a rehabilitation program focused on scar management, functional restoration, and symptom relief.
  Interventions: Device: ESWT Combined with Standard Rehabilitation
- Standard Rehabilitation Alone (Active Comparator): Participants assigned to this arm will receive the standard rehabilitation therapy protocol designed for post-burn scar management. This regimen includes physical, occupational, and scar-specific therapy sessions delivered in a standardized fashion without the addition of ESWT.
  Interventions: Behavioral: Standard Rehabilitation Therapy Alone

INTERVENTIONS:
Device: ESWT Combined with Standard Rehabilitation — Participants in the experimental arm will receive a combination intervention comprising ESWT delivered by certified technicians using a validated device for post-burn scars, along with standard rehabilitation therapy. ESWT sessions will be standardized (e.g., 3,000 pulses per session, weekly for 8 weeks) and will be integrated with a comprehensive rehabilitation program encompassing physical therapy, scar management exercises, and patient education. The specific parameters (e.g., energy level, frequency) will be reported based on established guidelines.
  Arms: ESWT Plus Standard Rehabilitation
Behavioral: Standard Rehabilitation Therapy Alone — Participants in the control arm will receive the institution's standard rehabilitation therapy for managing post-burn scars, including physical therapy, occupational therapy, and scar-massage techniques. Treatment frequency and duration will mirror the experimental arm's rehabilitation component to ensure consistency. No ESWT will be provided.
  Arms: Standard Rehabilitation Alone

SUMMARY:
This randomized controlled trial (RCT) will evaluate the cost-effectiveness of combining extracorporeal shock wave therapy (ESWT) with standard rehabilitation versus standard rehabilitation alone for the management of hypertrophic post-burn scars in adults. The study will assess clinical outcomes-such as pain intensity, pruritus, and scar quality-alongside economic outcomes including cost per quality-adjusted life year (QALY) gained, direct medical costs, and indirect costs (e.g., absenteeism and reduced productivity). Results will inform health policy and resource allocation decisions for advanced burn rehabilitation interventions.

DETAILED DESCRIPTION:
Post-burn hypertrophic scars can cause significant pain and pruritus, substantially affecting quality of life and functionality. Although ESWT has been recently associated with enhanced scar maturation and symptom reduction (Yang et al., 2022), its implementation into standard care is limited by a lack of economic evaluation. This trial is a prospective, randomized controlled study with an integrated cost-effectiveness analysis. Adult patients (aged 18-65) with hypertrophic scars at least 6 months post-burn injury will be recruited and stratified by scar severity. Participants will be randomized into one of two arms:

Arm 1 (Experimental): ESWT combined with standardized rehabilitation therapy. Arm 2 (Active Comparator): Standard rehabilitation therapy alone.

Primary clinical outcomes will include changes in pain intensity (measured on a Visual Analog Scale [VAS]), pruritus intensity (using the Itch Man Scale), and scar quality (assessed through the Vancouver Scar Scale [VSS]).

Economic outcomes will be determined by calculating the cost per QALY gained along with an assessment of both direct (therapy sessions, equipment use, hospital visits) and indirect costs (absenteeism, lost productivity).

Data will be collected at baseline and at follow-up visits at 1, 3, and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years. Documented hypertrophic scars following a burn injury, with scars present and stable for at least 6 months.

Moderate to severe scar severity as measured by a standardized clinical assessment.

Experiencing significant pain and/or pruritus related to the scar, with a baseline VAS score of ≥4.

Able to provide informed consent and comply with study procedures. Employed or engaged in daily activities such that indirect costs (absenteeism/reduced productivity) can be recorded.

Exclusion Criteria:

Pregnant or lactating women. Individuals with previous surgical scar revision or other invasive scar treatments within the last 6 months.

Patients with comorbid conditions (e.g., severe cardiovascular disease, uncontrolled diabetes) that could interfere with rehabilitation or ESWT.

Active skin infection in the area of the scar. Use of concurrent investigational therapies for scar management.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale [VAS]) | Assessed at baseline, 1 month, 3 months, and 6 months post-intervention.
  This measure evaluates the intensity of pain experienced by participants, using a 10-centimeter Visual Analog Scale where 0 indicates "no pain" and 10 indicates "worst pain imaginable." The VAS is a validated, standardized tool allowing for quantitative measurement of patient-reported pain intensity changes over time.
Cost per Quality-Adjusted Life Year (QALY) Gained | Evaluated at 6 months post-intervention.
  This economic outcome will be determined by calculating the incremental cost per QALY gained using validated health-related quality-of-life instruments (eg, EQ-5D) alongside hospital billing data. It compares the cumulative costs (both direct and indirect) and QALYs between the ESWT plus rehabilitation arm versus the rehabilitation alone arm over a 6-month period.

SECONDARY OUTCOMES:
Pruritus Intensity (Itch Man Scale) | Measured at baseline, 1 month, 3 months, and 6 months post-intervention.
  Pruritus will be quantified using the Itch Man Scale, a validated instrument designed to assess the severity and frequency of itching, which is a common symptom in post-burn scars.
Scar Quality (Vancouver Scar Scale [VSS]) | Assessed at baseline, 1 month, 3 months, and 6 months post-intervention.
  The Vancouver Scar Scale (VSS) will be employed to evaluate scar characteristics such as vascularity, pliability, height, and pigmentation. This scale is widely used for the objective assessment of burn scars.
Direct Medical Costs | Collated over the 6-month study period.
  Direct medical costs include expenditures for therapy sessions, ESWT equipment usage, hospital visits, and any additional medical services related to the intervention. Data will be extracted from hospital billing records.
Indirect Costs (Absenteeism and Reduced Productivity) | Evaluated cumulatively over the 6-month follow-up period.
  Indirect costs will encompass lost productivity and absenteeism, as estimated through participant-reported work absenteeism and validated economic questionnaires. These costs represent the broader societal impact of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No